CLINICAL TRIAL: NCT02399761
Title: Newborn Screening for Aromatic L-amino Acid Decarboxylase Deficiency
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201205084RIC
Record Dates: First submitted 2015-03-21; First posted 2015-03-26 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-10

CONDITIONS: Aromatic L-amino Acid Decarboxylase Deficiency
Keywords: AADC deficiency, newborn screening
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Parents of newborns will be invited to test if their newborns are affected with Aromatic L-amino Acid Decarboxylase (AADC) deficiency.

DETAILED DESCRIPTION:
Parents of newborns will be invited to test if their newborns are affected with Aromatic L-amino Acid Decarboxylase (AADC) deficiency. The routine newborn screening dried blood spots sample will be used to test if 3-O-methyldopa (3-OMD) concentration elevates. If positive of screening test, further confirmation tests including physical examination and for mutation. Genetic counseling and treatment option will be provided, too.

ELIGIBILITY:
Inclusion Criteria:

* Babies born in Taiwan receive regular new born screening suggested by Ministry of Heath and Welfare.
* Parents or Legal Guardian sign in the informed consent form.

Exclusion Criteria:

* Parents or Legal Guardian do not agree to sign in the informed consent form.

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborns whose parents agree to be tested
Sampling Method: Non-Probability Sample
Enrollment: 154795 (Actual)
Dates: Start 2012-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of newborns with AADC deficiency | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan